CLINICAL TRIAL: NCT04392336
Title: Development and Validation of a Feedback System for Tracking and Improving Trust/Respect in an Economically Disadvantaged Behavioral Health Population
Brief Title: Tracking and Improving Trust/Respect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Merakey Behavioral Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 830013
Record Dates: First submitted 2020-03-23; First posted 2020-05-18 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Impact of Feedback on Symptoms and Trust/Respect on Outcomes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trust/Respect feedback (Experimental): Clinicians with consumers in this arm receive feedback on trust/respect in addition to symptom feedback.
  Interventions: Other: Trust/Respect feedback
- No Trust/Respect feedback (No Intervention): Clinicians with consumers in this arm do not receive feedback on trust/respect and only receive symptom feedback.

INTERVENTIONS:
Other: Trust/Respect feedback — This feedback includes information on the level of trust/respect that a consumer has for their clinician in addition to symptom feedback.
  Arms: Trust/Respect feedback

SUMMARY:
This study will examine the efficacy of a feedback system for providers that tracks patient trust/respect on an ongoing basis and to test the hypothesis that receiving feedback on trust/respect will lead to improvements in patient satisfaction, functioning, symptoms, and trust/respect.

.

DETAILED DESCRIPTION:
This is a randomized effectiveness trial in which real-world providers will be given feedback on patient trust/respect. Approximately 40 clinicians, and up to 180 consumers will be enlisted participate in the randomized effectiveness trial. All enrolled patients will complete the BASIS-24, the Satisfaction with Care scale, and the Satisfaction with Social Roles and Activities Scale on handheld tablets or desktop computers at baseline. Patients will be randomized to one of two conditions. Patients in the first condition will attend therapy with clinicians who have received a standard automated outcome report, plus a report that contains information on the patient's trust/respect with suggestions for interventions if low/declining trust/respect is apparent. Patients in the second condition will attend therapy and complete the same measures as patients in the first condition, but their therapists will only receive a standard automated outcome report, without any patient information on trust/respect. At the time of the first therapy appointment and for all remaining therapy appointments, patients will complete four total measures: the new measure of trust/respect, the BASIS-24, the Satisfaction with Care scale, and the Satisfaction with Social Roles and Activities scale.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read at least at the 4th grade level
* 18 years of age and older
* Willingness to participate in research.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Change in PROMIS SF v2.0 scores | Up to 12 sessions, an average of 3 months
  Evaluates satisfaction with social roles and activities. Raw scores range from 4 to 20. This is a longitudinal assessment of change between multiple time points.

SECONDARY OUTCOMES:
Change in BASIS-24 scores | Up to 12 sessions, an average of 3 months
  The 24-item Behavior and Symptom Identification Scale is used to determine overall well-being. Scores range from 0 to 4. Lower scores indicate overall better well-being. This is a longitudinal assessment of change between multiple time points.
Change in Opinions about My Doctor/Therapist scores | Up to 12 sessions, an average of 3 months
  Asks participants questions regarding trust/respect for their clinician. Scores range from 1 to 7, with higher scores indicating greater trust/respect. This is a longitudinal assessment of change between multiple time points.
Change in Satisfaction with Care scores | Up to 12 sessions, an 3 months
  Evaluates satisfaction with care. Raw scores range from 1 to 7. This is a longitudinal assessment of change between multiple time points.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for data can be made through the PI.

REFERENCES:
- [Derived] Connolly Gibbons MB, Duong L, Zoupou E, Kashden J, Fisher J, Crits-Christoph P. Randomized controlled trial evaluating feedback to community-based therapists based on patient reports of trust and respect. J Consult Clin Psychol. 2023 Jun;91(6):337-349. doi: 10.1037/ccp0000807. Epub 2023 Mar 2. PMID 36862463